CLINICAL TRIAL: NCT04736706
Title: An Open-label, Randomized Phase 3 Study to Evaluate Efficacy and Safety of Pembrolizumab (MK-3475) in Combination With Belzutifan (MK-6482) and Lenvatinib (MK-7902), or MK-1308A in Combination With Lenvatinib, Versus Pembrolizumab and Lenvatinib, as First-Line Treatment in Participants With Advanced Clear Cell Renal Cell Carcinoma (ccRCC)
Brief Title: A Study of Pembrolizumab (MK-3475) in Combination With Belzutifan (MK-6482) and Lenvatinib (MK-7902), or Pembrolizumab/Quavonlimab (MK-1308A) in Combination With Lenvatinib, Versus Pembrolizumab and Lenvatinib, for Treatment of Advanced Clear Cell Renal Cell Carcinoma (MK-6482-012)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6482-012; MK-6482-012 (Other: MSD); jRCT2031210435 (Registry Identifier: jRCT(Japan Registry of Clinical Trials)); PHRR210911-003887 (Registry Identifier: Philippine Health Research Registry (PHRR)); 2020-002216-52 (EudraCT Number)
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Carcinoma, Renal Cell
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Hypoxia inducible factor (HIF); Hypoxia inducible factor 1B (HIF-1B); Hypoxia inducible factor 2 alpha (HIF-2 alpha)
MeSH Terms: conditions — Carcinoma, Renal Cell; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; belzutifan; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pembrolizumab + Belzutifan + Lenvatinib (Experimental): Participants will receive pembrolizumab 400 mg PLUS belzutifan 120 mg PLUS lenvatinib 20 mg. Pembrolizumab will be administered intravenously (IV) once every 6 weeks (Q6W) for up to 18 administrations (up to ~2 years). Belzutifan and lenvatinib will be administered orally once daily (QD) until progressive disease or discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Belzutifan; Drug: Lenvatinib
- Pembrolizumab/Quavonlimab + Lenvatinib (Experimental): Participants will receive pembrolizumab/quavonlimab (co-formulation of pembrolizumab 400 mg and quavonlimab 25 mg) PLUS lenvatinib 20 mg. Pembrolizumab/quavonlimab will be administered IV Q6W for up to 18 administrations (up to ~2 years). Lenvatinib will be administered orally QD until progressive disease or discontinuation.
  Interventions: Biological: Pembrolizumab/Quavonlimab; Drug: Lenvatinib
- Pembrolizumab + Lenvatinib (Active Comparator): Participants will receive pembrolizumab 400 mg PLUS lenvatinib 20 mg. Pembrolizumab will be administered IV Q6W for up to 18 administrations (up to ~2 years). Lenvatinib will be administered orally QD until progressive disease or discontinuation.
  Interventions: Biological: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Biological: Pembrolizumab — Pembrolizumab 400 mg administered Q6W via IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab + Belzutifan + Lenvatinib; Pembrolizumab + Lenvatinib
Drug: Belzutifan — Belzutifan 120 mg administered QD via oral tablet
  Other Names: MK-6482; PT2977; WELIREG™
  Arms: Pembrolizumab + Belzutifan + Lenvatinib
Biological: Pembrolizumab/Quavonlimab — Pembrolizumab/quavonlimab is a co-formulated product composed of pembrolizumab 400 mg in combination with quavonlimab 25 mg, administered Q6W via IV infusion
  Other Names: MK-1308A
  Arms: Pembrolizumab/Quavonlimab + Lenvatinib
Drug: Lenvatinib — Lenvatinib 20 mg administered QD via oral capsule
  Other Names: MK-7902; E7080; LENVIMA®

SUMMARY:
The goal of this study is to evaluate the efficacy and safety of pembrolizumab plus belzutifan plus lenvatinib or pembrolizumab/quavonlimab plus lenvatinib versus pembrolizumab plus lenvatinib as first-line treatment in participants with advanced clear cell renal cell carcinoma (ccRCC).

The primary hypotheses are (1) pembrolizumab plus belzutifan plus lenvatinib is superior to pembrolizumab plus lenvatinib with respect to progression-free survival (PFS) and overall survival (OS), in advanced ccRCC participants; and (2) pembrolizumab/quavonlimab plus lenvatinib is superior to pembrolizumab plus lenvatinib with respect to PFS and OS, in advanced ccRCC participants.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed diagnosis of RCC with clear cell component.
* Has received no prior systemic therapy for advanced ccRCC
* Male participants are abstinent from heterosexual intercourse or agree to use contraception during and for at least 7 days after last dose of study intervention with belzutifan and lenvatinib.
* Female participants are not pregnant or breastfeeding and are either not a woman of child-bearing potential (WOCBP) or use a contraceptive method that is highly effective or are abstinent from heterosexual intercourse during the intervention period and for at least 120 days after pembrolizumab or pembrolizumab/quavonlimab or for at least 30 days after last dose of lenvatinib or belzutifan, whichever occurs last
* Has adequately controlled blood pressure with or without antihypertensive medications
* Has adequate organ function.
* Participants receiving bone resorptive therapy must have therapy initiated at least 2 weeks prior to randomization/allocation

Exclusion Criteria:

* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has had major surgery, other than nephrectomy within 4 weeks prior to randomization
* Has known central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has received prior radiotherapy within 2 weeks prior to first dose of study intervention
* Has hypoxia or requires intermittent supplemental oxygen or requires chronic supplemental oxygen
* Has clinically significant cardiac disease within 12 months from first dose of study intervention
* Has a history of interstitial lung disease
* Has symptomatic pleural effusion; a participant who is clinically stable following treatment of this condition is eligible
* Has preexisting gastrointestinal or non-gastrointestinal fistula
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Has a known psychiatric or substance abuse disorder that would interfere with requirements of the study
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study drug; killed vaccines are allowed
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has a history of noninfectious pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of Hepatitis B
* Has radiographic evidence of intratumoral cavitation, encasement or invasion of a major blood vessel
* Has clinically significant history of bleeding within 3 months prior to randomization
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1653 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2026-10-29 (Estimated); Study Completion 2026-10-29 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 46 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR based on RECIST 1.1 will be presented.
Overall Survival (OS) | Up to approximately 66 months
  OS is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by BICR | Up to approximately 46 months
  ORR is defined as the percentage of participants who have a complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience a CR or PR as assessed by BICR based on RECIST 1.1 will be presented.
Duration of Response (DOR) Per RECIST 1.1 as Assessed by BICR | Up to approximately 66 months
  For participants who demonstrate a confirmed CR (disappearance of all target lesions) or confirmed PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until PD or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. The DOR as assessed by BICR based on RECIST 1.1 will be presented.
Number of Participants Who Experienced At least One Adverse Event (AE) | Up to approximately 66 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience at least one AE will be presented.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 66 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (262):
- United States (33):
  - The University of Alabama at Birmingham ( Site 0010), Birmingham, Alabama
  - UC San Diego ( Site 0050), La Jolla, California
  - Cedars Sinai Medical Center ( Site 0027), Los Angeles, California
  - University of California Irvine ( Site 0029), Orange, California
  - UCLA Hematology Oncology Santa Monica ( Site 0048), Santa Monica, California
  - Hartford Hospital ( Site 0024), Hartford, Connecticut
  - Advent Health Hematology & Oncology ( Site 0003), Orlando, Florida
  - University Cancer & Blood Center, LLC ( Site 0057), Athens, Georgia
  - Emory University Winship Cancer Institute ( Site 0012), Atlanta, Georgia
  - Rush University Medical Center ( Site 0040), Chicago, Illinois
  - Parkview Cancer Institute ( Site 0088), Fort Wayne, Indiana
  - Norton Cancer Institute - St. Matthews ( Site 0065), Louisville, Kentucky
  - Ochsner Medical Center ( Site 0049), New Orleans, Louisiana
  - New England Cancer Specialists ( Site 0082), Scarborough, Maine
  - Massachusetts General Hospital ( Site 0094), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center ( Site 0089), Boston, Massachusetts
  - Dana Farber Cancer Institute ( Site 0093), Boston, Massachusetts
  - Lahey Hospital & Medical Center ( Site 0090), Burlington, Massachusetts
  - Henry Ford Hospital ( Site 0038), Detroit, Michigan
  - Cancer & Hematology Centers of Western Michigan ( Site 0018), Grand Rapids, Michigan
  - HealthPartners Cancer Research Center-HealthPartners Frauenshuh Cancer Center ( Site 0005), Saint Louis Park, Minnesota
  - Regions Hospital ( Site 0095), Saint Paul, Minnesota
  - University of Mississippi Medical Center ( Site 0037), Jackson, Mississippi
  - Dartmouth Hitchcock Medical Center ( Site 0075), Lebanon, New Hampshire
  - Roswell Park Cancer Institute ( Site 0032), Buffalo, New York
  - R.J. Zuckerberg Cancer Center-Medical Oncology ( Site 0013), Lake Success, New York
  - Sidney Kimmel Center for Prostate and Urologic Cancers ( Site 0055), New York, New York
  - Oregon Health & Science University ( Site 0071), Portland, Oregon
  - Ralph H. Johnson VA Center ( Site 0073), Charleston, South Carolina
  - University of Tennessee Medical Center Knoxville ( Site 0019), Knoxville, Tennessee
  - Vanderbilt University Medical Center ( Site 0069), Nashville, Tennessee
  - UTSW Medical Center ( Site 0015), Dallas, Texas
  - Central Washington Health Services Association d/b/a Confluence Health ( Site 0061), Wenatchee, Washington
- Australia (5):
  - Liverpool Hospital ( Site 4006), Liverpool, New South Wales
  - Macquarie University ( Site 4007), Macquarie University, New South Wales
  - Lyell McEwin Hospital ( Site 4004), Elizabeth Vale, South Australia
  - Monash Health ( Site 4008), Clayton, Victoria
  - Fiona Stanley Hospital ( Site 4009), Murdock, Western Australia
- Brazil (8):
  - Oncocentro Ceara ( Site 0309), Fortaleza, Ceará
  - Centro de Pesquisas Clinicas em Oncologia ( Site 0306), Cachoeiro de Itapemirim, Espírito Santo
  - Centro Avançado de Tratamento Oncológico- CENATRON-Clinical Research ( Site 0303), Belo Horizonte, Minas Gerais
  - Liga Norte Riograndense Contra o Cancer ( Site 0308), Natal, Rio Grande do Norte
  - Hospital de Clinicas de Porto Alegre ( Site 0310), Porto Alegre, Rio Grande do Sul
  - Instituto do Cancer do Estado de Sao Paulo - ICESP ( Site 0302), São Paulo
  - BP - A Beneficencia Portuguesa de São Paulo-Medical Oncology ( Site 0300), São Paulo
  - A.C. Camargo Cancer Center ( Site 0301), São Paulo
- Canada (5):
  - Tom Baker Cancer Centre ( Site 0119), Calgary, Alberta
  - BC Cancer - Vancouver Center ( Site 0120), Vancouver, British Columbia
  - Hamilton Health Sciences-Juravinski Cancer Centre ( Site 0117), Hamilton, Ontario
  - Sunnybrook Research Institute ( Site 0116), Toronto, Ontario
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 0, Québec, Quebec
- Chile (5):
  - IC La Serena Research ( Site 0403), La Serena, Coquimbo Region
  - Servicios Medicos Urumed ( Site 0405), Rancagua, Lbtdr Gen Bernardo O Higgins
  - Fundacion Arturo Lopez Perez ( Site 0400), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 0401), Santiago, Region M. de Santiago
  - Centro Investigacion Cancer James Lind ( Site 0402), Temuco, Región de la Araucanía
- China (30):
  - The First Afflilated Hospital of Bengbu Medical College-Urology Surgery ( Site 6041), Bengbu, Anhui
  - Cancer Hospital Chinese Academy of Medical Science-Oncology ( Site 6026), Beijing, Beijing Municipality
  - Peking University First Hospital ( Site 6011), Beijing, Beijing Municipality
  - Beijing Cancer hospital-Renal carcinoma and melanoma ( Site 6000), Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital ( Site 6009), Chongqing, Chongqing Municipality
  - The First Affiliated Hospital Of Fujian Medical University-Urology ( Site 6038), Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University-Urology ( Site 6001), Xiamen, Fujian
  - SUN YAT-SEN UNIVERSITY CANCER CENTRE ( Site 6003), Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University-Urology ( Site 6036), Guangzhou, Guangdong
  - Guangzhou First People's Hospital ( Site 6007), Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University-Urology Surgery ( Site 6005), Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital-urology ( Site 6015), Harbin, Heilongjiang
  - Henan Cancer Hospital-Urology ( Site 6006), Zhengzhou, Henan
  - Wuhan Union Hospital ( Site 6002), Wuhan, Hubei
  - Xiangya Hospital Central South University ( Site 6034), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 6020), Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School-Urology ( S, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University-Urology ( Site 6025), Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University ( Site 6019), Nanchang, Jiangxi
  - Jiangxi Provincial Cancer Hospital ( Site 6042), Nanchang, Jiangxi
  - The First Affiliated Hospital of Xi'an Jiaotong University ( Site 6014), Xi'an, Shaanxi
  - Renji Hospital Shanghai Jiao Tong University School of Medicine ( Site 6017), Shanghai, Shanghai Municipality
  - Shanghai Tenth People's Hospital ( Site 6023), Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University-Urology Surgery ( Site 6016), Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital ( Site 6029), Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical University ( Site 6032), Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University ( Site 6024), Hangzhou, Zhejiang
  - The First Hospital of Jiaxing ( Site 6033), Jiaxing, Zhejiang
  - Ningbo First Hospital-Urology ( Site 6028), Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University-Urology Surgery ( Site 6021), Wenzhou, Zhejiang
- Colombia (7):
  - Instituto de Cancerología S.A Clínica de las Americas (ICCLA) ( Site 0500), Medellín, Antioquia
  - Clinica de la Costa S.A.S. ( Site 0502), Barranquilla, Atlántico
  - Administradora Country SA - Clinica del Country ( Site 0504), Bogotá, Bogota D.C.
  - Instituto Nacional de Cancerología E.S.E. ( Site 0503), Bogotá, Bogota D.C.
  - Sociedad de Oncología Y Hematología del Cesar S.A.S. ( Site 0505), Valledupar, Cesar Department
  - Oncólogos del Occidente S.A ( Site 0501), Pereira, Risaralda Department
  - Fundacion Cardiovascular de Colombia ( Site 0506), Piedecuesta, Santander Department
- Croatia (3):
  - Klinicki Bolnicki Centar Zagreb ( Site 3200), Zagreb, City of Zagreb
  - Klinički Bolnički Centar Split ( Site 3202), Split, Split-Dalmatia County
  - Klinicki bolnicki centar "Sestre milosrdnice" ( Site 3201), Zagreb, Zagreb County
- Czechia (7):
  - Masarykuv onkologicky ustav ( Site 2203), Brno, Brno-mesto
  - Nemocnice AGEL Novy Jicin a.s. ( Site 2202), Nový Jičín, Moravskoslezský kraj
  - Fakultni nemocnice Ostrava ( Site 2208), Ostrava, Moravskoslezský kraj
  - Fakultni nemocnice u sv. Anny v Brne ( Site 2205), Brno, South Moravian
  - Fakultni nemocnice Olomouc ( Site 2200), Olomouc
  - Fakultni Thomayerova nemocnice ( Site 2201), Prague
  - 2 LF UK a FN Motol ( Site 2207), Prague
- Denmark (2):
  - Herlev Hospital ( Site 1700), Herlev, Capital Region
  - Odense University Hospital ( Site 1701), Odense, Region Syddanmark
- Finland (4):
  - Kuopion Yliopistollinen Sairaala ( Site 1803), Kuopio, Northern Savonia
  - TAYS ( Site 1801), Tampere, Pirkanmaa
  - TYKS ( Site 1802), Turku, Southwest Finland
  - HYKS ( Site 1800), Helsinki, Uusimaa
- France (9):
  - Institut Paoli Calmettes ( Site 1206), Marseille, Bouches-du-Rhone
  - CHU Jean Minjoz ( Site 1205), Besançon, Doubs
  - Institut Claudius Regaud ( Site 1214), Toulouse, Haute-Garonne
  - Clinique Francois Chenieux ( Site 1209), Limoges, Haute-Vienne
  - Clinique Ambroise Pare Beuvry ( Site 1213), Beuvry, Hauts-de-France
  - CHU Angers ( Site 1200), Angers, Maine-et-Loire
  - CH Lyon Sud Hospices Civils de Lyon ( Site 1203), Pierre-Bénite, Rhone
  - Gustave Roussy ( Site 1207), Villejuif, Val-de-Marne
  - Hopital Tenon ( Site 1212), Paris
- Germany (3):
  - Universitaetsklinik fuer Urologie ( Site 1300), Tübingen, Baden-Wurttemberg
  - Helios Kliniken Schwerin GmbH ( Site 1302), Schwerin, Mecklenburg-Vorpommern
  - Charite Universitaetsmedizin Berlin ( Site 1301), Berlin
- Guatemala (6):
  - Centro Medico Integral de Cancerologia CEMIC ( Site 0701), Salcajá, Departamento de Quetzaltenango
  - Oncomedica ( Site 0700), Guatemala City
  - Grupo Angeles SA ( Site 0705), Guatemala City
  - Sanatorio Nuestra Senora del Pilar ( Site 0702), Guatemala City
  - Medi-K Cayala ( Site 0703), Guatemala City
  - Centro Regional de Sub Especialidades Medicas SA ( Site 0704), Quetzaltenango
- Hungary (6):
  - Bekes Megyei Kozponti Korhaz - Pandy Kalman Tagkorhaza ( Site 2309), Gyula, Bekes County
  - Bacs-Kiskun Megyei Korhaz-Onkoradiologiai Kozpont ( Site 2308), Kecskemét, Bács-Kiskun county
  - Jász-Nagykun-Szolnok Vármegyei Hetényi Géza Kórház ( Site 2300), Szolnok, Jász-Nagykun-Szolnok
  - Markusovszky Egyetemi Oktatokorhaz ( Site 2303), Szombathely, Vas County
  - Orszagos Onkologiai Intezet ( Site 2304), Budapest
  - Debreceni Egyetem Klinikai Kozpont ( Site 2301), Debrecen
- Ireland (2):
  - Beaumont Hospital ( Site 6101), Dublin
  - Tallaght University Hospital ( Site 6100), Dublin
- Italy (7):
  - Azienda Ospedaliero - Universitaria Policlinico di Modena ( Site 1404), Modena, Emilia-Romagna
  - Ospedale San Raffaele-Oncologia Medica ( Site 1417), Milan, Lombardy
  - Fondazione Policlinico Universitario A. Gemelli ( Site 1414), Rome, Roma
  - Azienda Ospedaliera Policlinico di Bari ( Site 1411), Bari
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 1409), Milan
  - Istituto Nazionale Tumori Fondazione Pascale ( Site 1412), Napoli
  - Azienda Ospedaliera S. Maria di Terni ( Site 1410), Terni
- Japan (23):
  - Fujita Health University ( Site 5003), Toyoake, Aichi-ken
  - Chiba cancer center ( Site 5021), Chiba, Chiba
  - National Cancer Center Hospital East ( Site 5000), Kashiwa, Chiba
  - Ehime University Hospital ( Site 5020), Tōon, Ehime
  - Sapporo Medical University Hospital ( Site 5008), Sapporo, Hokkaido
  - Hokkaido University Hospital ( Site 5013), Sapporo, Hokkaido
  - Kanagawa cancer center ( Site 5016), Yokohama, Kanagawa
  - Nara Medical University Hospital ( Site 5002), Kashihara, Nara
  - Kindai University Hospital- Osakasayama Campus-Urology ( Site 5010), Sayama, Osaka
  - Osaka University Hospital ( Site 5012), Suita, Osaka
  - Saitama Medical University International Medical Center ( Site 5015), Hidaka, Saitama
  - Hamamatsu University School of Medicine University Hospital ( Site 5004), Hamamatsu, Shizuoka
  - Tokyo Medical And Dental University Medical Hospital-Urology ( Site 5009), Bunkyō, Tokyo
  - Toranomon Hospital ( Site 5001), Minato-ku, Tokyo
  - Toyama University Hospital ( Site 5014), Toyoma, Toyama
  - Kyushu University Hospital ( Site 5005), Fukuoka
  - Kumamoto University ( Site 5022), Kumamoto
  - Niigata University Medical & Dental Hospital ( Site 5024), Niigata
  - Okayama University Hospital ( Site 5017), Okayama
  - Tokushima University Hospital-Department of Urology ( Site 5019), Tokushima
  - Nippon Medical School Hospital ( Site 5006), Tokyo
  - Tokyo Women's Medical University Adachi Medical Center ( Site 5023), Tokyo
  - Keio university hospital ( Site 5011), Tokyo
- Malaysia (4):
  - Hospital Sultan Ismail ( Site 4303), Johor Bahru, Johor
  - Institut Kanser Negara - National Cancer Institute ( Site 4302), Putrajaya, Putrajaya
  - Hospital Kuala Lumpur ( Site 4301), Kuala Lumpur
  - Universiti Malaya Medical Centre ( Site 4300), Kuala Lumpur
- Mexico (5):
  - Hospital Civil de Guadalajara Fray Antonio Alcalde ( Site 0610), Guadalajara, Jalisco
  - Instituto Nacional de Cancerologia ( Site 0602), Mexico City, Mexico City
  - I CAN Oncology SA de SV ( Site 0601), Monterrey, Nuevo León
  - Hospital H+ Queretaro-Cuidados Oncológicos ( Site 0608), Querétaro City, Querétaro
  - Centro de Investigacion Clinica de Oaxaca ( Site 0605), Oaxaca City
- Norway (6):
  - Akershus universitetssykehus ( Site 2000), Lorenskog, Akershus
  - Soerlandet sykehus HF Kristiansand ( Site 2007), Kristiansand, Aust-Agder
  - Helse Bergen HF - Haukeland Universitetssykehus ( Site 2002), Bergen, Hordaland
  - St. Olavs Hospital HF ( Site 2005), Trondheim, Sor-Trondelag
  - Oslo Universitetssykehus Radiumhospitalet ( Site 2001), Oslo
  - Sykehuset Østfold HF Kalnes ( Site 2003), Grålum, Østfold fylke
- Philippines (3):
  - Manila Doctors Hospital ( Site 4601), Manila, National Capital Region
  - The Medical City ( Site 4602), Pasig, National Capital Region
  - Cardinal Santos Medical Center ( Site 4603), San Juan City, National Capital Region
- Poland (7):
  - Przychodnia Lekarska KOMED ( Site 2419), Konin, Greater Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny w Poznaniu ( Site 2406), Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 2420), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Radomskie Centrum Onkologii ( Site 2418), Radom, Masovian Voivodeship
  - Luxmed Onkologia sp. z o. o. ( Site 2412), Warsaw, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie ( Site 2405), Warsaw, Masovian Voivodeship
  - Szpital Wojewodzki im. Mikolaja Kopernika ( Site 2407), Koszalin, West Pomeranian Voivodeship
- Romania (4):
  - Spitalul Judetean de Urgenta Alba Iulia ( Site 2502), Alba Iulia, Alba
  - S.C. Centrul de Oncologie Sf. Nectarie SRL ( Site 2501), Craiova, Dolj
  - Policlinica Oncomed SRL ( Site 2506), Timișoara, Timiș County
  - S.C.Focus Lab Plus S.R.L ( Site 2503), Bucharest
- Russia (9):
  - Altay Regional Oncology Dispensary ( Site 2610), Barnaul, Altayskiy Kray
  - Ivanovo Regional Oncology Dispensary ( Site 2615), Ivanovo, Ivanovo Oblast
  - Krasnoyarsk Regional Clinical Oncological Dispensary ( Site 2609), Krasnoyarsk, Krasnoyarsk Krai
  - The Loginov Moscow Clinical Scientific Center ( Site 2604), Moscow, Moscow
  - Moscow Oncological Clinical Dispensary #1 ( Site 2619), Moscow, Moscow
  - FBHI Privolzhsky District Medical Center of the FMBA ( Site 2611), Nizhny Novgorod, Nizhny Novgorod Oblast
  - Nizhniy Novgorod Region Oncology Dispensary ( Site 2621), Nizhny Novgorod, Nizhny Novgorod Oblast
  - Scientific Research Oncology Institute n.a. N.N.Petrov ( Site 2617), Saint Petersburg, Sankt-Peterburg
  - City clinical oncological dispensary ( Site 2605), Saint Petersburg, Sankt-Peterburg
- Serbia (3):
  - Klinicki centar Srbije. ( Site 3333), Belgrade, Beograd
  - Klinicki centar Nis ( Site 3322), Niš, Nisavski Okrug
  - Institut za onkologiju Vojvodine ( Site 3311), Kamenitz, Sremski Okrug
- South Africa (10):
  - Cancer Care Langenhoven Drive Oncology Centre ( Site 3009), Port Elizabeth, Eastern Cape
  - Wits Clinical Research ( Site 3012), Johannesburg, Gauteng
  - Sandton Oncology Medical Group PTY LTD ( Site 3000), Johannesburg, Gauteng
  - Univ. Pretoria and Steve Biko Academic Hospitals ( Site 3002), Pretoria, Gauteng
  - Life Wilgers Hospital ( Site 3004), Pretoria, Gauteng
  - Mary Potter Oncology Centre, Little Company of Mary Hospital ( Site 3001), Pretoria, Gauteng
  - Vaal Triangle Oncology Centre ( Site 3010), Vereeniging, Gauteng
  - Groote Schuur Hospital ( Site 3011), Cape Town, Western Cape
  - Cape Town Oncology Trials Pty Ltd ( Site 3006), Kraaifontein, Western Cape
  - Cancercare Rondebosch Oncology ( Site 3005), Rondebosch, Western Cape
- South Korea (7):
  - National Cancer Center ( Site 4202), Goyang-si, Kyonggi-do
  - Chungnam National University Hospital ( Site 4205), Daejeon, Taejon-Kwangyokshi
  - Korea University Anam Hospital ( Site 4206), Seoul
  - Seoul National University Hospital ( Site 4201), Seoul
  - Severance Hospital Yonsei University Health System ( Site 4204), Seoul
  - Asan Medical Center ( Site 4203), Seoul
  - Samsung Medical Center ( Site 4200), Seoul
- Spain (6):
  - Instituto Catalan de Oncologia - ICO ( Site 1502), L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marques de Valdecilla ( Site 1501), Santander, Cantabria
  - Institut Català d'Oncologia (ICO) - Girona ( Site 1500), Girona, Gerona
  - Hospital Clinico San Carlos ( Site 1503), Madrid
  - Hospital Universitario 12 de Octubre ( Site 1505), Madrid
  - Hospital Universitario Virgen de la Victoria ( Site 1504), Málaga
- Sweden (5):
  - Lanssjukhuset Ryhov ( Site 2103), Jönköping, Jönköping County
  - Karolinska Universitetssjukhuset Solna ( Site 2100), Stockholm, Stockholm County
  - Akademiska Sjukhuset ( Site 2105), Uppsala, Uppsala County
  - Norrlands Universitetssjukhus ( Site 2106), Umeå, Västerbotten County
  - Sahlgrenska Universitetssjukhuset ( Site 2102), Gothenburg, Västra Götaland County
- Taiwan (6):
  - Chang Gung Medical Foundation. Kaohsiung Branch ( Site 4405), Kaohsiung City
  - Taichung Veterans General Hospital ( Site 4403), Taichung
  - National Cheng Kung University Hospital ( Site 4404), Tainan
  - National Taiwan University Hospital ( Site 4401), Taipei
  - Taipei Veterans General Hospital ( Site 4402), Taipei
  - Chang Gung Medical Foundation-Linkou Branch-Urology ( Site 4406), Taoyuan District
- Thailand (2):
  - Ramathibodi Hospital. ( Site 4500), Bangkok, Bangkok
  - Siriraj Hospital ( Site 4501), Bangkok, Bangkok
- Turkey (Türkiye) (7):
  - Ankara Universitesi Tip Fakultesi ( Site 2902), Ankara
  - Hacettepe Universitesi Tıp Fakultesi ( Site 2903), Ankara
  - Trakya University Medical Faculty Balkan Oncology Hospital ( Site 2906), Edirne
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi ( Site 2900), Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 2901), Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi ( Site 2904), Izmir
  - Dokuz Eylul Universitesi Tip Fakultesi Hastanesi ( Site 2905), Izmir
- Ukraine (10):
  - Cherkasy Regional Oncology Dispensary ( Site 2704), Cherkasy, Cherkasy Oblast
  - Chernihiv Medical Center of Modern Oncology ( Site 2709), Chernihiv, Chernihiv Oblast
  - Clinical oncology dispensary of Dnipro ( Site 2700), Dnipro, Dnipropetrovsk Oblast
  - ME І.І. Mechnykov Dnipro Regional Clinical Hospital ( Site 2710), Dnipropetrovsk, Dnipropetrovsk Oblast
  - Ivano-Frankivsk Regional Hospital-Urology department ( Site 2707), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Ivano-Frankivsk Regional Oncology Clinical Dispensary ( Site 2711), Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Regional Oncology Center of Kharkiv ( Site 2708), Kharkiv, Kharkivs’ka Oblast’
  - Reg. Clinical Center of Urology and Nephrology n.a. V. I. Shapoval ( Site 2715), Kharkiv, Kharkivs’ka Oblast’
  - Kyiv City Clinical Oncology Center ( Site 2706), Kyiv, Kyivska Oblast
  - Lviv State Regional Oncological Center ( Site 2712), Lviv, Lviv Oblast
- United Kingdom (3):
  - Addenbrookes Hospital ( Site 3110), Cambridge, Cambridgeshire
  - Barts Health NHS Trust - St Bartholomew s Hospital ( Site 3116), London, England
  - Mount Vernon Cancer Centre ( Site 3101), Northwood, London, City of

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Choueiri TK, Powles T, Voss MH, Plimack ER, Gurney H, Song Y, Perini RF, Rodriguez-Lopez K, Rini BI. LITESPARK-012: pembrolizumab plus lenvatinib with or without belzutifan or quavonlimab for advanced renal cell carcinoma. Future Oncol. 2023 Dec;19(40):2631-2640. doi: 10.2217/fon-2023-0283. Epub 2023 Oct 26. PMID 37882432
- [Derived] Ged Y, Markowski MC, Singla N, Rowe SP. The shifting treatment paradigm of metastatic renal cell carcinoma. Nat Rev Urol. 2022 Nov;19(11):631-632. doi: 10.1038/s41585-022-00651-9. PMID 36064785
- See also: Merck Clinical Trials Information — https://merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26235&tenant=MT_MSD_9011